CLINICAL TRIAL: NCT00112411
Title: Dose-ranging Double-blind, Placebo-controlled Efficacy Comparison of Two Bronchodilator Inhalers in Pediatric Asthmatics
Brief Title: Comparison of Two Bronchodilator Inhalers in Pediatric Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IXR-204-25-167
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Bronchodilator Agents

INTERVENTIONS:
Drug: Bronchodilator

SUMMARY:
This study is designed to evaluate the single-dose effectiveness of two bronchodilator inhalers given at two dose levels in pediatric asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma for a minimum of six months duration that has been stable for at least four weeks
* Predicted FEV1 60-90%
* Demonstration of 12% airway reversibility

Exclusion Criteria:

* Continuous requirement for beta-blockers, monoamine oxidase (MAO) inhibitors, tricyclic antidepressants, anticholinergics and/or steroids other than those inhaled;
* Presence of clinically-significant non-asthmatic acute or chronic disease

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-06-30 (Actual); Primary Completion 2005-09-30 (Actual); Study Completion 2005-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Allergy Associates Medical Group, Inc., San Diego, California
  - Aeroallergy Research Labs of Savannah, Inc., Savannah, Georgia
  - University of Louisville, Louisville, Kentucky
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Mississippi Asthma and Allergy Clinic, Jackson, Mississippi
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Medical Research Network, The Woodlands, Texas